CLINICAL TRIAL: NCT07274735
Title: Combined Effect Of Intraneural Facilitation Therapy And Otago Exercise On Pain, Balance And Quality Of Life In Patients With Diabetic Peripheral Neuropathy
Brief Title: Combined Effects of INF and OEP in Patients With Diabetic Peripheral Neuropathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0269 Rameen Shahzad
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic Nephropathies; Exercise; Musculoskeletal Manipulations; Peripheral Neuropathy; Quality of Life
MeSH Terms: conditions — Diabetic Nephropathies; Motor Activity; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intraneural facilitation therapy (Experimental): The intervention will consist of 24 sessions delivered three times per week over eight weeks, with each session lasting 50-60 minutes. Effects will be measured at baseline (before treatment), after the 4th week and after 8th week (post treatment)
  Interventions: Other: Intraneural facilitation therapy
- Otago exercise program (Experimental): Otago exercise training was conducted 3 times a week for a total of 50 min per session, including 5 min of warm-up and 5 min of cool-down. Effects will be measured at baseline, at 4th weeks and at 8th week. The exercises consisted of the following strengthening exercises: knee extensors, knee flexors, hip abductors, ankle plantar flexors, and ankle dorsiflexors. The balance retraining exercises consisted of the following: knee bends, backwards walking, walking and turning around, sideways walking, tandem stance, tandem walk, one leg stand, heel walking, toe walking, heel toe walking backwards, and sit to stand
  Interventions: Other: Otago exercise program
- Intraneural facilitation therapy with Otago exercise program (Experimental): The exercise intervention will be an 8 week, 3xweek, and 50-60 min class following the 20-30min OEP curriculum with 20-30 min /sessions of intraneural facilitation therapy per week. Effects will be measured at baseline, at 4th weeks and at 8th week
  Interventions: Other: Intraneural facilitation therapy with Otago exercise program

INTERVENTIONS:
Other: Intraneural facilitation therapy — The intervention will consist of 24 sessions delivered three times per week over eight weeks, with each session lasting 50-60 minutes. Effects will be measured at baseline (before treatment), after the 4th week and after 8th week (post treatment)
  Arms: Intraneural facilitation therapy
Other: Otago exercise program — Otago exercise training was conducted 3 times a week for a total of 50 min per session, including 5 min of warm-up and 5 min of cool-down. Effects will be measured at baseline, at 4th weeks and at 8th week. The exercises consisted of the following strengthening exercises: knee extensors, knee flexors, hip abductors, ankle plantar flexors, and ankle dorsiflexors. The balance retraining exercises consisted of the following: knee bends, backwards walking, walking and turning around, sideways walking, tandem stance, tandem walk, one leg stand, heel walking, toe walking, heel toe walking backwards, and sit to stand
  Arms: Otago exercise program
Other: Intraneural facilitation therapy with Otago exercise program — The exercise intervention will be an 8 week, 3xweek, and 50-60 min class following the 20-30min OEP curriculum with 20-30 min /sessions of intraneural facilitation therapy per week. Effects will be measured at baseline, at 4th weeks and at 8th week
  Arms: Intraneural facilitation therapy with Otago exercise program

SUMMARY:
DPN often leads to balance issues, sensory deficits, and chronic pain, which can severely impact daily functioning and independence. INF therapy aims to improve nerve blood flow and alleviate neuropathic symptoms through manual techniques, while the Otago Exercise Program focuses on enhancing strength and balance to reduce fall risk. By comparing these two interventions, this study seeks to identify effective strategies that can improve balance, reduce pain, and enhance the quality of life for individuals suffering from DPN

DETAILED DESCRIPTION:
This study addresses a gap in existing literature by comparing the effects of intraneural facilitation therapy and Otago exercise in improving balance, pain and QOL among DPN patients. While both Intraneural Facilitation (INF) therapy and the Otago Exercise Program have been acknowledged for their individual benefits, their comparative effectiveness in the context of diabetic peripheral neuropathy (DPN) has not been adequately explored. This study aims to bridge this gap by examining which intervention more effectively improves quality of life, reduces pain, and enhances balance in DPN patients, thus providing essential insights for optimizing treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75years
* Both male and female patients will be included in the study
* Patient with type 2 diabetes mellitus (diagnosed by the physician)
* Patients with a score ≥ 4 on DN4 scale
* Patients have a score on the Timed Up-and-Go (TUG) test of less than 15 s
* Able to walk at least 10 meters long

Exclusion Criteria:

* Patient with presence of any other systemic disease rather than diabetes such as end-stage renal failure, uncontrolled hypertension, severe dyslipidemia, chronic liver disease, autoimmune disease, advanced chronic obstructive pulmonary disease etc
* Patients with documented active alcohol or drug misuse
* Patient with total or partial amputation of lower extremities
* Participants will be also excluded if they were morbidly obese or if pregnant (self-reported)
* Patient with active inflammations or other inflammatory neuropathies including chronic inflammatory demyelinating polyneuropathy, proximal diabetic neuropathy, chemotherapy-induced peripheral neuropathy, autonomic neuropathies, or other neuropathies not associated with DM such as B12 deficiency

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-01-17 (Estimated); Study Completion 2026-01-17 (Estimated)

PRIMARY OUTCOMES:
DN4 | 8th week
  The DN4 Questionnaire is a screening tool for neuropathic pain consisting of 10 interview questions (DN4-interview) and physical tests which has been validated for the diagnosis of diabetic peripheral neuropathy in western populations. The DN4 questionnaire is used to screen for the presence of neuropathic pain. This questionnaire consisted of 4 sections; 3 sections concerned with symptoms review and associated symptoms and the 4th section reserved for physical examination.
Mini BESTest scale | 8th week
  The Mini-BESTest has 14 items, scored from 0-2, so the maximum score is 28
Quality of Life- Diabetic Neuropathy Questionnaire | 8th week
  It is an extensive and validated 35-item questionnaire that has been developed to encompass the complete range of Diabetic Neuropathy (DN) symptoms associated with small fiber, large fiber, and autonomic neuropathy. It is composed of two sections: one focusing on the symptoms experienced by diabetic patients and the other on how the patient's neuropathy affects their activities of daily living (ADLs).

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | 8th week
  Numeric Pain Rating Scale is a subjective measure 11 point (0-10) numerical scale which is a commonly used outcome measure to assess pain intensity, including in patients with diabetic peripheral neuropathy. Its score ranges from 0 indicating no pain at all to 10 indicating worst pain
TUG test | 8th week
  In this test, participants are asked to stand up from a chair, walk 3 m, turn, walk 3 m back and sit down again. The time taken to perform this task indicates high or low falls risk. The cut-off scores reported in the articles varied from 10.9 s to 13 s.
Ankle brachial index (ABI) | 8th week
  ABI (Osc-ABI) during the first measurement by the first observer were 89.1%, 94.4%, 94.1%, 91.8%, and 92.4%, sensitivity and specificity respectively normal value will be 0.9-1.4, higher: greater than 1.4, typically indicative of vessel stiffening. Low: less than 0.9 means narrowing of vessels, non-measurable: unable to occlude blood vessel at 300mmHG of pressure application

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (1):
- Rasheed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker NA, Vuong D, Bussell M, Gharibvand L, Lee S, Tsao B. Prospective, Randomized, Double-Blinded, Sham-Controlled Pilot Study of Intraneural Facilitation as a Treatment for Carpal Tunnel Syndrome. Arch Rehabil Res Clin Transl. 2022 Mar 29;4(2):100193. doi: 10.1016/j.arrct.2022.100193. eCollection 2022 Jun. PMID 35756982
- [Background] Alnajafi KZ-S. The Impact of Intraneural Facilitation Therapy on Diabetic Peripheral Neuropathy. 2021.
- [Background] Kadir MI, Hardiyanty N, Adliah F. A pilot study of the effect of otago exercise program on fall risk and quality of life of older women. Physical Therapy Journal of Indonesia. 2021;2(1):1-4.
- [Background] Jahanpeyma P, Kayhan Kocak FO, Yildirim Y, Sahin S, Senuzun Aykar F. Effects of the Otago exercise program on falls, balance, and physical performance in older nursing home residents with high fall risk: a randomized controlled trial. Eur Geriatr Med. 2021 Feb;12(1):107-115. doi: 10.1007/s41999-020-00403-1. Epub 2020 Nov 25. PMID 33237565
- [Background] Brown JJ, Colberg SR, Pribesh S, Baskette KG, Vinik AI. A comparison of neuropathy quality of life tools: Norfolk QOL-DN, PN-QOL-97, and NeuroQOL-28. Medical Research Archives. 2021;9(11)
- [Background] Agoons BB, Tchapmi D, Boli AO, Katte J-C. Clinical utility of the DN4 questionnaire in the assessment of neuropathic pain in patients with type 2 diabetes: Experience from a newly-created diabetes clinic in Cameroon. PAMJ-Clinical Medicine. 2020;3(165).
- [Background] Lytras D, Sykaras E, Iakovidis P, Komisopoulos C, Chasapis G, Mouratidou C. Effects of a modified Otago exercise program delivered through outpatient physical therapy to community-dwelling older adult fallers in Greece during the COVID-19 pandemic: a controlled, randomized, multicenter trial. Eur Geriatr Med. 2022 Aug;13(4):893-906. doi: 10.1007/s41999-022-00656-y. Epub 2022 May 24. PMID 35606677
- [Background] Spallone V, Morganti R, D'Amato C, Greco C, Cacciotti L, Marfia GA. Validation of DN4 as a screening tool for neuropathic pain in painful diabetic polyneuropathy. Diabet Med. 2012 May;29(5):578-85. doi: 10.1111/j.1464-5491.2011.03500.x. PMID 22023377
- [Background] Shakya BM, Shrestha A, Poudyal AK, Shrestha N, Acharya B, Gurung R, et al. Nepalese version of Douleur Neuropathique 4 (DN4) questionnaire for Assessment of Neuropathic pain: A Validation Study. medRxiv. 2021:2021.09. 17.21263734.
- [Background] Zielinski J, Morawska-Kochman M, Zatonski T. Pain assessment and management in children in the postoperative period: A review of the most commonly used postoperative pain assessment tools, new diagnostic methods and the latest guidelines for postoperative pain therapy in children. Adv Clin Exp Med. 2020 Mar;29(3):365-374. doi: 10.17219/acem/112600. PMID 32129952
- [Background] Vinik EJ, Hayes RP, Oglesby A, Bastyr E, Barlow P, Ford-Molvik SL, Vinik AI. The development and validation of the Norfolk QOL-DN, a new measure of patients' perception of the effects of diabetes and diabetic neuropathy. Diabetes Technol Ther. 2005 Jun;7(3):497-508. doi: 10.1089/dia.2005.7.497. PMID 15929681
- [Background] Alghamdi M, Owolabi LF, Adamu B, Taura MG, Jibo A, Almansour M, Alaklabi SN, Alghamdi MA, Imam IA, Abdelrazak R, Rafaat A, Aliyu MH. Disease-specific quality of life in patients with diabetic neuropathy. Saudi Med J. 2022 Apr;43(4):408-417. doi: 10.15537/smj.2022.43.4.20210861. PMID 35414620
- [Background] Smith SC, Lamping DL, Maclaine GD. Measuring health-related quality of life in diabetic peripheral neuropathy: a systematic review. Diabetes Res Clin Pract. 2012 Jun;96(3):261-70. doi: 10.1016/j.diabres.2011.11.013. Epub 2011 Dec 10. PMID 22154463
- [Background] King L, Horak F. On the mini-BESTest: scoring and the reporting of total scores. Phys Ther. 2013 Apr;93(4):571-5. doi: 10.2522/ptj.2013.93.4.571. No abstract available. PMID 23547173
- [Background] Yingyongyudha A, Saengsirisuwan V, Panichaporn W, Boonsinsukh R. The Mini-Balance Evaluation Systems Test (Mini-BESTest) Demonstrates Higher Accuracy in Identifying Older Adult Participants With History of Falls Than Do the BESTest, Berg Balance Scale, or Timed Up and Go Test. J Geriatr Phys Ther. 2016 Apr-Jun;39(2):64-70. doi: 10.1519/JPT.0000000000000050. PMID 25794308
- [Background] Meekes WM, Korevaar JC, Leemrijse CJ, van de Goor IA. Practical and validated tool to assess falls risk in the primary care setting: a systematic review. BMJ Open. 2021 Sep 29;11(9):e045431. doi: 10.1136/bmjopen-2020-045431. PMID 34588228
- [Background] Ichihashi S, Desormais I, Hashimoto T, Magne J, Kichikawa K, Aboyans V. Accuracy and Reliability of the Ankle Brachial Index Measurement Using a Multicuff Oscillometric Device Versus the Doppler Method. Eur J Vasc Endovasc Surg. 2020 Sep;60(3):462-468. doi: 10.1016/j.ejvs.2020.06.013. Epub 2020 Aug 3. PMID 32763120
- [Background] Leem SH, Kim JH, Lee BH. Effects of Otago exercise combined with action observation training on balance and gait in the old people. J Exerc Rehabil. 2019 Dec 31;15(6):848-854. doi: 10.12965/jer.1938720.360. eCollection 2019 Dec. PMID 31938708